CLINICAL TRIAL: NCT01598545
Title: Determination of the ED50 of Intrathecal Hydromorphone for Post-cesarean Section Pain Relief
Brief Title: Hydromorphone and C-section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Grant Lynde, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00058097
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydromorphone (Experimental): Laboring patients having a cesarean section will receive ED50 of hydromorphone one time intrathecally
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone will be administered one time intrathecally to laboring patients to determine the ED50 for pain relief.

SUMMARY:
This study will investigate the dose of hydromorphone which will relieve the pain of women following a cesarean section when delivered directly in the area around the spinal cord (i.e., intrathecal injection). The primary objective is to determine the dose of intrathecal hydromorphone that results in a pain score of less than 3 out of 10 12 hours after intrathecal injection in 50% of women. Secondary objectives include determining the average amount of time patients obtain pain relief after injection. Other secondary objectives include determining the frequency and severity of side-effects associated with intrathecal administration of hydromorphone, including: bradycardia, hypotension, respiratory depression, apnea, pruritus, rash, nausea, vomiting, and drowsiness. Thirty women admitted to labor and delivery for planned cesarean section desiring will be consented for the study. The starting dose of intrathecal hydromorphone will be 6 mcg. The up-and-down sequential allocation method of statistical analysis will be used, meaning that each subsequent dose will be dependent upon the result obtained from the prior dose - ergo, if the initial subject has pain relief, the second subject will receive 4 mcg (2 mcg less), but if the initial subject does not have pain relief, the second subject will receive 8 mcg (2 mcg more) of hydromorphone.

After the intrathecal injection is given, patients will undergo their cesarean section. The patient's pain will be assessed at 6, 12, and 18 hours post-injection using a questionnaire. The patient's medical record will be reviewed to determine when she first requested supplemental pain medication. A pain score of less than three will be a positive result. A pain score of three or greater will be a negative result. Blood pressure, heart rate, arterial oxygen saturation, 5 and 10 minute APGAR scores, and any side effects will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women undergoing cesarean section

Exclusion Criteria:

* Any comorbidities other than obesity, hypertension, fetal anomalies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant C Lynde, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled from January 2013 to June 2014 at Grady Memorial Hospital.
Groups:
- Hydromorphone: Laboring patients having a cesarean section will receive ED50 of hydromorphone one time intrathecally
  Hydromorphone: Hydromorphone will be administered one time intrathecally to laboring patients to determine the ED50 for pain relief.
  ED50 of hydromorphone was 5.6 mcg +/- 1.8 mcg.
Period: Overall Study
Arm/Group | Hydromorphone
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores, Visual Analogue Pain Scale
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: 12 hours after intrathecal injection
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 2.75 [0 to 8]

2. Secondary Outcome: Pain Scores, Visual Analogue Pain Scale
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: Baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 0.45 [0 to 4]

3. Secondary Outcome: Pain Scores, Visual Analogue Pain Scale
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: 6 hours after intrathecal injection
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 4.4 [0 to 10]

4. Secondary Outcome: Pain Scores, Visual Analogue Pain Scale
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: 18 hours after intrathecal injection
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 3.05 [0 to 8]

5. Secondary Outcome: Pain Scores, Visual Analogue Pain Scale
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: 24 hours after intrathecal injection
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 3.3 [0 to 7]

ADVERSE EVENTS:
Groups:
- Hydromorphone: Laboring patients receive ED50 of hydromorphone one time intrathecally
  Hydromorphone: Hydromorphone will be administered one time intrathecally to laboring patients to determine the ED50 for pain relief.
  ED50 of hydromorphone was 5.6 mcg +/- 1.8 mcg.
Arm/Group | Hydromorphone
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes